CLINICAL TRIAL: NCT06103760
Title: Positioning of Esketamine Treatment in the Real-world Management of Depression
Acronym: PoET
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Collaborators: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Principal Investigator, Gin Malhi, Professor, Royal North Shore Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/PID01587
Record Dates: First submitted 2023-10-15; First posted 2023-10-27 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants with Major Depressive Disorder (Other): Intranasal esketamine to be self-administered by participants under direct supervision of a healthcare professional. First initial dose is 56mg and subsequent doses will be 56mg or 84mg. Esketamine will be administered twice weekly for weeks 1-4, once weekly for weeks 5-8, and once weekly/once fortnightly/once monthly as clinically indicated for weeks 9-25. After each treatment phase, participants will be re-assessed through a comprehensive battery of assessments and dose adjustments will be performed by the study psychiatrist base on tolerability, treatment response, and ongoing consent.
  Interventions: Drug: Esketamine Nasal Spray [Spravato]

INTERVENTIONS:
Drug: Esketamine Nasal Spray [Spravato] — This is an uncontrolled, single arm, naturalistic study. There will be three treatment phases: Phase 1 - Acute treatment phase (weeks 1-4); Phase 2 - Maintenance treatment phase (weeks 5-8); Phase 3 - Continuation treatment phase (Weeks 9-25). Phase 1 is the critical component of our study as it determines our primary outcomes.
  Other Names: Spravato

SUMMARY:
The goal of this naturalistic, open label, single arm intervention study is to investigate the effects of Esketamine in treating depression.The main aims to answer are:

* to investigate whether Esketamine is effective when added to ongoing antidepressant treatment
* to identify patient characteristics that will determine a therapeutic response to Esketamine in real-world practice

Participants will:

* attend the clinic for supervised self-administration of intranasal Esketamine treatment
* be observed for 2 hours following Esketamine administration including blood pressure monitoring
* be asked to complete a battery of questionnaires
* be reimbursed for travel expenses

DETAILED DESCRIPTION:
Depression is a common mental illness, and it is one of the leading causes of disease burden worldwide. Fortunately, there are many effective treatments available for depression, including lifestyle changes, psychological treatments, and medications such as antidepressants. However, not all patients will respond to the first treatment prescribed. Some patients may only experience a 'partial response', where a few treatments help their depression somewhat, but they do not achieve a full recovery. Currently, the reasons why some patients do not respond, or only experience a partial response to an antidepressant, is not fully understood.

Recently, researchers have been investigating new medications that may help patients recover from depression. One of these new medications is Esketamine, which is a relatively new molecule derived from a drug called Ketamine - an anaesthetic that has been used medically for decades. Researchers have been investigating the antidepressant properties of Ketamine for a long time. It is thought that Ketamine, and its derivative, Esketamine, help to treat depression for a number of reasons. However, it is not yet known which patients benefit most from Esketamine when used in conjunction with conventional antidepressants. In addition, we do not yet understand how the effect of Esketamine is impacted by other treatments that a patient may be taking for their depression. Finally, it has not yet been investigated how patients with a partial response to an antidepressant will benefit from adding Esketamine to their therapeutic regimen without switching to a new baseline antidepressant. Therefore, there are two principle aims of this study 1) to investigate whether Esketamine is effective when added to ongoing antidepressant treatment and 2) to identify patient characteristics that will determine a therapeutic response to Esketamine in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-65 years old
2. Diagnosis of Major Depressive Disorder (MDD)
3. Currently depressed
4. Had an inadequate response to 2 or more courses of antidepressants (of adequate dose and duration)
5. Be maintained on their current antidepressant medication or psychological therapy at the time of enmrolment
6. Able to understand and provide informed consent

Exclusion Criteria:

1. Concurrent diagnoses:

   * Participants with other 'Diagnostic and Statistical Manual of Mental Disorders' (DSM-5) e.g., current substance misuse disorder, bipolar disorder, schizophrenia
   * Participants who are unable to understand the study and therefore unable to provide informed consent
2. Pregnancy:

   * Participants who are pregnant and/or breastfeeding
   * Participants who are not willing to avoid pregnancy for themselves or their partners during the study by using effective birth control methods
3. Current medications:

   * Participants taking a total daily dose of benzodiazepines greater than the equivalent of 6mg/day of lorazepam
   * Participants on complementary and alternative medicine therapies i.e., St John's wort, Chinese medicines, and various herbal and homeopathic treatments
4. Stimulants

   * Participants taking stimulants such as methylphenidate, amphetamine, and dextroamphetamine for a diagnosis such as ADHD can still have Esketamine provided they do not continue taking stimulants concurrently for the duration of the study.
   * Concurrent use is excluded due to the synergistic effect with Esketamine that can cause increased blood pressure.
5. Medical history:

   * Participants with current or past history of seizures (uncomplicated childhood febrile seizures with no sequelae are not exclusionary)
   * Participants with a history of uncontrolled hypertension
   * Participants with uncontrolled diabetes mellitus
   * Participants with aneurysmal vascular disease including thoracic and abdominal aorta, intracranial and peripheral arterial vessels, or arteriovenous malformation, intracerebral haemorrhage
   * Participants with untreated glaucoma, current penetrating or perforating eye injury, brain injury, hypertensive encephalopathy, intrathecal therapy with ventricular shunts, or any other condition associated with increased intracranial pressure or increased intraocular pressure or planned eye surgery
   * Participants who are currently receiving electroconvulsive therapy (ECT) or have received ECT in the past month.
6. Substance Misuse History:

   * Participants who have ever had a substance misuse disorder involving any of the following over their lifetime: ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3,4-methylenedioxy-methamphetamine (MDMA), or other hallucinogen use history
   * Participants with hypersensitivity to Esketamine, Ketamine, or any of the excipients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of treatment responders determined by a 50% reduction on the Hamilton Depression Rating Scale (HAM-D) 17-Item scoring. | At the end of week 4
  Hamilton Depression Rating Scale (HAM-D) 17-Item scoring
Mean depression score on the Quick Inventory of Depressive Symptomatology Self-report (QIDS-SR) 16-Item. | Baseline, at the end of weeks 1,2,3, and 4 (primary time point); and further after week 8 and week 12 after Esketamine was commenced.
  Quick Inventory of Depressive Symptomatology Self-report (QIDS-SR) 16-Item.
Global functioning determined by Clinical Global Impression (CGI) score. | Baseline, week 1, week 2, week 3, week 4 (primary time point), week 8 and week 12 after Esketamine was commenced.
  Clinical Global Impression (CGI)

SECONDARY OUTCOMES:
Change in mood symptom scores assessed using the visual analogue scale (self-reported) | Baseline, after treatment day 1 and day 3 of each week until Esketamine is ceased.
  Visual analogue scale (self-reported)
Depressive symptoms assessed using the Beck Depression Inventory (BDI) 21-Item. | Baseline and at week 4 after Esketamine was commenced.
  Beck Depression Inventory (BDI) 21-Item.
Anxiety symptoms assessed using the State-Trait Anxiety Inventory (STAI) | Baseline and at week 4 after Esketamine was commenced.
  State-Trait Anxiety Inventory (STAI)

CONTACTS AND LOCATIONS:
Overall Officials: Gin Malhi, Principal Investigator — Royal North Shore Hospital, University of Sydney
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No